CLINICAL TRIAL: NCT05290337
Title: Phase 2 Study of Zanubrutinib Plus RCHOP (ZR-CHOP) in Newly Diagnosed Diffuse Large B-cell Lymphoma With Specific Gene Abnormality
Brief Title: ZR-CHOP in DLBCL With Specific Gene Abnormality
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junning Cao, MD, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZIDEA
Record Dates: First submitted 2022-02-10; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Zanubrutinib; gene mutation; MYC translocation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZR-CHOP (Experimental)
  Interventions: Drug: zanubrutinib

INTERVENTIONS:
Drug: zanubrutinib — BTK inhibitor

SUMMARY:
This is a phase 2, single center clinical trial. to evaluating the efficacy and safety of Zanubrutinib in combination with R-CHOP in newly diagnosed diffuse large B-cell lymphoma with specific gene abnormality.

DETAILED DESCRIPTION:
This is a phase 2, single center clinical trial. to evaluating the efficacy and safety of Zanubrutinib in combination with R-CHOP in newly diagnosed diffuse large B-cell lymphoma with specific gene abnormality, including MYC translocation, MYD88 mutation, CD79B mutation, NOTCH1 mutation and TP53 mutation. all patients received 6 cycle therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. histological confirmed, newly-diagnosed diffuse large B-cell lymphoma with one of the following gene abnormality including MYC translocation, MYD88 mutation, CD79B mutation, NOTCH1 mutation and TP53 mutation;
3. Eastern Cooperative Oncology Group (ECOG) status of 0-1; 4) hospitalized patients and received the whole cycle treatment in Fudan University Shanghai Cancer Center-
4. normal hematological, hepatic and renal function.
5. Life expectancy of more than 3 months;
6. Patients had at least one measurable target lesion;
7. LVEF ≥ 50%
8. signed informed consent forms

Exclusion Criteria:

1. hypersensitivity to immunoglobulin;
2. primary central nerves lymphoma
3. History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix;
4. With contraindication of steroid including uncontrolled diabetes;
5. Serious uncontrolled diseases and intercurrent infection;
6. Pregnant or lactating women;
7. hepatitis B infection with HBV-DNA ≥ 104

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-01-04 (Estimated); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
3-year progression free survival | assessed up to 36 months
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Objective response rate | assessed up to 36 months
  complete remission and partial remission
3-year event free survival | assessed up to 36 months
  From date of enrollment until the date of an event, including progression, death from any cause, new treatment.
3-year overall survival | assessed up to 36 months
  From date of enrollment until the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No